CLINICAL TRIAL: NCT02739321
Title: A Randomized, Cross-Over Study of the Efficacy of Mattress Technology in Improving the Sleep Quality of Children With ASD and Sleep Disturbances
Brief Title: Examining the Efficacy of Mattress Technology in Improving the Sleep Quality of Children With ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Kugona LLC (Unknown)
Responsible Party: Principal Investigator, Thomas W. Frazier, Ph.D, Thomas W. Frazier, Ph.D, The Cleveland Clinic
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 14-066
Record Dates: First submitted 2014-07-21; First posted 2016-04-15 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Autism Spectrum Disorders
Keywords: Autism; ASD; Sleep; Mattress
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mattress Technology On then Off (Experimental): Intervention: Sound to Sleep System will be turned on for the first two weeks of the study allowing the participant sleeping atop the mattress to feel the vibrations synced to the audio input. Sound to sleep system will be turned on during this phase of the study. The sound to sleep system will sync an audio input with the vibrations of the mattress technology and allow the user to control the intensity of the vibration.
  No intervention: The mattress technology will be turned off for the second two weeks of the study. During this time, there will be no intervention.
  Interventions: Device: Sound to Sleep System
- Mattress Technology Turned Off then On (Experimental): No intervention: For the first two weeks of the study, the mattress technology will not be turned off. There will be no intervention during this time.
  Intervention: Sound to Sleep System will be turned on for the second two weeks of the study allowing the participant sleeping atop the mattress to feel the vibrations synced to the audio input. Sound to sleep system will be turned on during this phase of the study. The sound to sleep system will sync an audio input with the vibrations of the mattress technology and allow the user to control the intensity of the vibration.
  Interventions: Device: Sound to Sleep System

INTERVENTIONS:
Device: Sound to Sleep System — Sound to Sleep System is a minimal risk device that is embedded in a mattress boxspring. The device syncs with an audio input and emits tactile vibrations in sync with the audio input.

SUMMARY:
The purpose of the present study is to evaluate the tolerability and efficacy of the Sound To Sleep System™ in improving the sleep quality of children with Autism Spectrum Disorder (ASD). The Sound To Sleep System™ is a mattress foundation designed to improve sleep quality in individuals with ASD and sleep disturbance by providing mattress vibrations that accompany and sync with auditory stimulation. For the present study, the primary objectives are as follows:

* Study Aim 1 - To determine whether the use of the Sound To Sleep System™ in ASD-affected children with sleep disturbances is well tolerated as defined by group drop-out proportion due to issues with the mattress technology.

The study will also explore the following objectives:

* Study Aim 2 - To determine the efficacy of the Sound To Sleep System™ in improving sleep quality as measured by parent reported sleep quality in ASD-affected children with sleep disturbances. (Please note Study Aim 2 was changed from clinician-rated to parent-rated because we were not able to collect clinician-rated sleep quality information).
* Study Aim 3 - To determine the tolerability of the Sound To Sleep System™ as defined by study drop-out due to any reason and caregiver ratings of ease of mattress technology use.
* Study Aim 4 - To determine whether use of the mattress technology improves functioning as defined by secondary outcome measures.

DETAILED DESCRIPTION:
The present study aims to evaluate the tolerability and efficacy of a new mattress technology in improving the sleep quality of children with Autism Spectrum Disorder (ASD). Clinical and population studies indicate that children with ASD exhibit elevated rates of sleep disturbance compared to their typically-developing peers and that 50% to 80% of children with ASD have sleep problems. Sleep disturbance can include bedtime resistance, sleep onset latency, nighttime awakenings, decreased total sleep time, early morning awakenings, and other measures of sleep quality. Sleep problems in children with ASD are associated with greater externalizing and internalizing behavior problems during the waking day, poorer adaptive functioning, and can cause significant parental stress. Previous studies have examined the effectiveness of behavioral treatments, environmental modifications, melatonin, and psychopharmacologic treatments in decreasing the rates of sleep disturbance. However, none of these approaches have identified treatments that are effective for all ASD-affected children with sleep difficulties. Given the high prevalence of sleep disturbance in this population, there is a great need to identify additional treatments that may improve sleep in children with ASD.

The purpose of the present study is to evaluate the tolerability and efficacy of the Sound To Sleep System™ using a single blind (actigraphy scoring blinded), cross-over design. The Sound To Sleep System™ is a mattress foundation designed to improve sleep quality in individuals with ASD and sleep disturbance by providing mattress vibrations that accompany and sync with auditory stimulation. For the present study, the primary objectives are as follows:

Study Aim 1- To determine whether the use of the Sound To Sleep System™ in ASD-affected children with sleep disturbances is well tolerated as defined by group drop-out proportion due to issues with the mattress technology.

The study will also explore the following objectives:

Study Aim 2- To determine the efficacy of the Sound To Sleep System™ in improving parent-reported sleep quality in ASD-affected children with sleep disturbances.

Study Aim 3- To determine the tolerability of the Sound To Sleep System™ as defined by study drop-out due to any reason and caregiver ratings of ease of mattress technology use.

Study Aim 4- To determine whether use of the mattress technology improves functioning as defined by secondary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* ASD Diagnosis
* 2.5-12.99 Years of Age
* Sleep Difficulty as indicated by significant sleep disturbance on the Child Sleep Habits Questionnaire
* If participant is using medication or attends therapy, it must be stable four (4) weeks prior to their study participation and throughout the 5-6 week study period.

Exclusion Criteria:

* Age less than 2.5 years or more than 12.99 years
* Individuals who may have medication or therapy changes 4 weeks prior to study start date or during the study period
* An participant diagnosed with epilepsy, Fragile X, Downs Syndrome, seizure disorder, Neurofibromatosis, or Tuberous Sclerosis
* Any child with a pacemaker or other electrical device

Ages: 30 Months to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2014-05; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Frazier, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Center for Autism, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrolled participants take part in a one-week lead in period during which time all participants sleep with the box spring foundation of the new mattress technology, but with the mattress technology turned off, and wear an actigraphy watch. Participants who are unable to tolerate the actigraphy watch or the box spring foundation are excluded.
Groups:
- Mattress Technology On Then Off: Intervention: The mattress technology is turned on allowing the participant sleeping atop the mattress to feel the vibrations synced to the audio input.
  Sound to Sleep System turned on: For the first two weeks of the study, the sound to sleep system will be turned on during this arm of the study. For the second two weeks of the study, the Sound to Sleep System will be turned off, there is no intervention.
- Mattress Technology Turned Off Then On: Intervention: The mattress technology is turned on allowing the participant sleeping atop the mattress to feel the vibrations synced to the audio input.
  Sound to Sleep System: For the first two weeks of the study, the Sound to Sleep System is turned off, there is no intervention. For the second two weeks of the study, the Sound to Sleep System is turned on.
Period: Overall Study
Arm/Group | Mattress Technology On Then Off | Mattress Technology Turned Off Then On
Started | 23 | 22
Completed | 20 | 18
Not Completed | 3 | 4
Not completed — Lack of Efficacy | 1 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Mattress Technology On: Intervention: The first two weeks of the study the mattress technology will be turned on allowing the participant sleeping atop the mattress to feel the vibrations synced to the audio input. The second two weeks of the study, the mattress technology will be turned off, there will be no intervention.
  Sound to Sleep System turned on: The first two weeks of the study the sound to sleep system will be turned on during this arm of the study. The second two weeks of the study, the sound to sleep system will be turned off, there will be no intervention.
- Mattress Technology Turned Off: Intervention: The first two weeks of the study there will be no intervention. The second two weeks of the study, the mattress technology will be turned on allowing the participant sleeping atop the mattress to feel the vibrations synced to the audio input.
  Sound to Sleep System: The first two weeks of the study the sound to sleep system will be turned off, there will be no intervention. The second two weeks of the study the sound to sleep system will be turn on.
- Total: Total of all reporting groups
Arm/Group | Mattress Technology On | Mattress Technology Turned Off | Total
Number analyzed (Participants) | 23 | 22 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23 | 22 | 45
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.0 (2.5) | 6.2 (2.8) | 6.1 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 19 | 17 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 21 | 21 | 42
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 22 | 45

OUTCOME MEASURES:

1. Primary Outcome: Compare Percentage of Participants Who Drop Out of Study as a Measure of Toleration of Mattress Technology
Description: Compare percentage of drop-out, in this cohort, due to issues with the mattress technology (e.g. ease of use, inability to fall asleep) to a population expected drop-out rate of 30% using a one-sample proportion test.
Time Frame: up to 6 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Mattress Technology On Then Off: For the first two weeks of the study, the mattress technology is turned on
  For the second two weeks of the study, the mattress technology is turned off, there is no intervention.
  Intervention: The mattress technology is turned on allowing the participant sleeping atop the mattress to feel the vibrations synced to the audio input.
- Mattress Technology Off Then On: For the first two weeks of the study, the mattress technology is turned off, there is no intervention.
  For the second two weeks of the study, the mattress technology is turned on
  Intervention: The mattress technology is turned on allowing the participant sleeping atop the mattress to feel the vibrations synced to the audio input.
Arm/Group | Mattress Technology On Then Off | Mattress Technology Off Then On
Number analyzed (Participants) | 23 | 22
Participants | 1 | 1
Statistical Analysis 1: Comparison: Mattress Technology On Then Off vs Mattress Technology Off Then On; Test type: Non-Inferiority — Hypothesized benchmark of 30%; p < .001, t-test, 2 sided; Risk Difference (RD) = 25.6

2. Secondary Outcome: Parent Reported Quality of Sleep Across Treatment Conditions
Description: Within subjects comparison of the average daily, parent reported sleep quality across on and off conditions using a Likert-type scale of 1-7 in which 1 is "extremely poor" and 7 is "exceptional"
Time Frame: Average daily score, across up to 2 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Mattress Technology On: Participants who slept with the mattress technology turned on in either the first or second two weeks of the study.
- Mattres Technology Off: Participants who slept with the mattress technology turned off in either the first or second two weeks of the study.
Arm/Group | Mattress Technology On | Mattres Technology Off
Number analyzed (Participants) | 45 | 45
units on a scale | 4.9 [4.67 to 5.14] | 4.3 [4.05 to 4.54]
Statistical Analysis 1: Comparison: Mattress Technology On vs Mattres Technology Off; Test type: Superiority; p = .001, Mixed Models Analysis

3. Secondary Outcome: Total Time Asleep Recorded by Actigraphy Watch
Description: Within subjects comparison of the average total sleep time (hours) in the on and off conditions as recorded by actigraphy watch
Time Frame: Average of daily measure, across up to 2 weeks
Measure: Mean (Standard Error); unit: Hours
Groups:
- Mattress Technology Off: Participants who slept with the mattress technology turned off in either the first or second two weeks of the study.
Arm/Group | Mattress Technology On | Mattress Technology Off
Number analyzed (Participants) | 45 | 45
Hours | 8.35 (0.22) | 7.99 (0.22)
Statistical Analysis 1: Comparison: Mattress Technology On vs Mattress Technology Off; Test type: Superiority; p = 0.001, Mixed Models Analysis; Mean Difference (Final Values) = .12

4. Secondary Outcome: Total Time to Fall Asleep (Sleep Latency) Recorded by Actigraphy Watch
Description: Within subjects comparison of sleep latency (minutes) recorded by actigraphy watch in the on and off conditions
Time Frame: Average of daily measure, across up to 2 weeks
Measure: Mean (Standard Error); unit: Minutes
Arm/Group | Mattress Technology On | Mattress Technology Off
Number analyzed (Participants) | 45 | 45
Minutes | 14.11 (5.75) | 18.20 (6)
Statistical Analysis 1: Comparison: Mattress Technology On vs Mattress Technology Off; Test type: Superiority; p = .268, Mixed Models Analysis; Median Difference (Final Values) = 4.09

5. Secondary Outcome: Total Time Awake During Night Recorded by Actigraphy Watch
Description: Within subjects comparison of total time awake during night (minutes) recorded by actigraphy watch in both on and off conditions
Time Frame: Average of daily measure, across up to 2 weeks
Measure: Mean (Standard Error); unit: Minutes
Arm/Group | Mattress Technology On | Mattress Technology Off
Number analyzed (Participants) | 45 | 45
Minutes | 17.85 (0.92) | 18.79 (0.93)
Statistical Analysis 1: Comparison: Mattress Technology On vs Mattress Technology Off; Test type: Superiority; p = .058, Mixed Models Analysis; Mean Difference (Final Values) = 0.94

6. Secondary Outcome: Percentage of Time in Bed That the Participant Spent Sleeping (Sleep Efficiency) Recorded by Actigraphy Watch.
Description: Within subjects comparison of time spent sleeping (sleep efficiency as percentage) recorded by actigraphy in both the one and off conditions.
Time Frame: Average of daily measure, across up to 2 weeks
Measure: Mean (Standard Error); unit: percentage of time
Arm/Group | Mattress Technology On | Mattress Technology Off
Number analyzed (Participants) | 45 | 45
percentage of time | 78.27 (1.48) | 75.45 (1.38)
Statistical Analysis 1: Comparison: Mattress Technology On vs Mattress Technology Off; Test type: Superiority; p = .001, Mixed Models Analysis; Mean Difference (Final Values) = 2.82

7. Secondary Outcome: Caregiver-Rated Severity of Social Deficits as Measured by the Social Responsiveness Scale 2 (SRS-2)
Description: Within subjects comparison of average Social Responsiveness Scale -2 (SRS-2) T-scores in baseline, and on and off conditions.
  SRS-2 T-score ranges from 30-90 (M = 50, SD = 10). Higher T-scores indicate a greater extent of social communication deficits.
Time Frame: Baseline, 2 weeks, 4 weeks
Measure: Mean (Standard Error); unit: T-score
Groups:
- Baseline: All participants before they were randomized into arms
Arm/Group | Baseline | Mattress Technology On | Mattress Technology Off
Number analyzed (Participants) | 45 | 45 | 45
T-score | 76.40 (1.61) | 73.68 (1.72) | 74.77 (1.71)
Statistical Analysis 1: Comparison: Mattress Technology On vs Mattress Technology Off; Test type: Superiority; p = .232, Mixed Models Analysis

8. Secondary Outcome: Caregiver-Rated Severity Problem Behaviors as Measured by the Aberrant Behavior Checklist (ABC)
Description: Within subjects comparison of the parent completed Aberrant Behavior Checklist (ABC) total raw score in the baseline, and on and off conditions.
  The ABC measures the level of challenging behavior of individuals in and across 5 subdomains (Irritability, lethargy, stereotypy, hyperactivity, inappropriate speech) using a Likert-type scale of 0-3 in which 0 is "not at all a problem" and 3 is "the problem is severe in degree". The sum raw scores of these subdomains make up the total ABC raw score (range = 0-174) in which a higher score indicates more severe challenging behaviors.
Time Frame: Baseline, 2 weeks, 4 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Baseline | Mattress Technology On | Mattress Technology Off
Number analyzed (Participants) | 45 | 45 | 45
units on a scale | 56.9 (4.25) | 48.61 (4.96) | 55.37 (4.91)
Statistical Analysis 1: Comparison: Mattress Technology On vs Mattress Technology Off; Test type: Superiority; p = 0.100, Mixed Models Analysis

9. Secondary Outcome: Caregiver-Rated Communication Problems as Measured by the CCC-2
Description: Within subjects comparison of the average Children's Communication Checklist (CCC-2) General Communication Composite standard scores across baseline, and on and off conditions.
  CCC-2 is a parent questionnaire that assesses children's communication skills across 10 domains using a 4-point Likert type scale (0=less than once a week/never to 3=several times a day/always). The general communication composite standard score based on age norms was used to asses overall communication competency (M=100, SD=15). Lower general communication composite scores indicate a higher likelihood of significant communication problems.
Time Frame: Baseline, 2 weeks, 4 weeks
Measure: Mean (Standard Error); unit: Standard Score
Groups:
- Mattress Technonlogy Off: Participants who slept with the mattress technology turned off in either the first or second two weeks of the study.
Arm/Group | Baseline | Mattress Technology On | Mattress Technonlogy Off
Number analyzed (Participants) | 45 | 45 | 45
Standard Score | 48.31 (2.59) | 52.31 (2.79) | 50.79 (2.74)
Statistical Analysis 1: Comparison: Mattress Technology On vs Mattress Technonlogy Off; Test type: Superiority; p = 0.285, Mixed Models Analysis

10. Secondary Outcome: Caregiver-Rated Problems With Sleep Habits as Measured by the FISH
Description: Within subjects comparison of the Family Inventory of Sleep Hygiene (FISH) average total raw scores across baseline, and on and off conditions.
  The FISH is a parent-completed questionnaire that assesses sleep hygiene-related behaviors in children using a 5-point Likert scale (1=Never, 2=occasionally, 3=Sometimes, 4=Usually, 5=Always). Typically parents rate these behaviors with reference to the past month, but for the present study they were asked to rate for only the previous two weeks to correspond to each mattress condition. The total raw score was used to asses sleep hygiene (Range = 12-60, in which higher scores are indicative of better sleep hygiene-related behaviors).
Time Frame: Baseline, 2 weeks, 4 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Baseline | Mattress Technology On | Mattress Technology Off
Number analyzed (Participants) | 45 | 45 | 45
units on a scale | 46.82 (0.70) | 48.79 (0.89) | 47.15 (0.88)
Statistical Analysis 1: Comparison: Mattress Technology On vs Mattress Technology Off; Test type: Superiority; p = 0.089, Mixed Models Analysis

11. Secondary Outcome: Caregiver-Rated Sleep Disturbance as Measured by the Children's Sleep Habits Questionnaire (CSHQ)
Description: Within subjects comparison of the Children's Sleep Habits Questionnaire CSHQ average total raw scores across baseline and on and off conditions.
  The CSHQ is a parent-completed questionnaire that measures a variety of sleep-related problems using a 3-point Likert-scale (1=rarely/0 to 1 times per week, 2= sometimes/2-4 times per week, 3=usually/5-7 times per week). Ordinarily, parents rate these behaviors for the pas week but for the present study they were instructed to rate for the past two weeks to correspond to the mattress on and off conditions. The total raw scores were use to evaluate overall sleep difficulties (Range = 45-135, in which a higher score is indicative of more sleep problems).
Time Frame: Baseline, 2 weeks, 4 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Baseline | Mattress Technology On | Mattress Technology Off
Number analyzed (Participants) | 45 | 45 | 45
units on a scale | 56.53 (1.11) | 49.13 (1.37) | 52.66 (1.35)
Statistical Analysis 1: Comparison: Mattress Technology On vs Mattress Technology Off; Test type: Superiority; p = 0.040, Mixed Models Analysis

12. Secondary Outcome: Caregiver-Rated Sensory Issues Across Domains as Measured by the SSPQ
Description: Within subjects comparison of the Short Sensory Profile Questionnaire (SSPQ) average total raw scores across baseline and on and off conditions.
  The SSPQ is a parent-completed questionnaire that measures behaviors related to sensory processing abnormalities. Items are based on a 5-point Liker scale ranging from 1=always to 5=never. The total raw score was used to evaluate overall sensory abnormalities (Range=38-190). Lower scores indicate a higher probability of sensory processing abnormalities.
Time Frame: Baseline, 2 weeks, 4 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Baseline | Mattress Technology On | Mattress Technology Off
Number analyzed (Participants) | 45 | 45 | 45
units on a scale | 124.58 (3.14) | 129.43 (4.02) | 125.49 (3.98)
Statistical Analysis 1: Comparison: Mattress Technology On vs Mattress Technology Off; Test type: Superiority; p = 0.471, Mixed Models Analysis

13. Secondary Outcome: Caregiver-Rated of Quality of Life as Measured by the CFQL-2 Questionnaire
Description: Within subjects comparison of the Child and Family Quality of Life 2 (CFQL-2), quality of life average total raw scores across baseline and on and off conditions.
  The CFQL-2 is a parent questionnaire that evaluation seven different aspects of child and family quality of life (child, family, caregiver, financial, partner relationship, external support, and coping quality of life). An adapted version was used that decreased the number of total items from 32 to 26 and added an additional item to each scale to specifically evaluate changes of the past two weeks in quality of life. Items use a 5-point Likert scale ranging from (1=strongly disagree/decreased substantially to 3=neutral/same to 5=strongly agree/improved substantially). The total raw score was used to evaluate overall quality of life for child and family (Range=26-130). A lower, overall score indicates a lower quality of life for the child and their family.
Time Frame: Baseline, 2 weeks, 4 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Baseline | Mattress Technology On | Mattress Technology Off
Number analyzed (Participants) | 45 | 45 | 45
units on a scale | 79.95 (1.77) | 84.54 (2.19) | 79.87 (2.14)
Statistical Analysis 1: Comparison: Mattress Technology On vs Mattress Technology Off; Test type: Superiority; p = 0.015, Mixed Models Analysis

14. Secondary Outcome: Caregiver-Rated Measure of Challenging Behavior/Task Compliance as Measured by the Daily Sleep Diary
Description: Within subjects comparison of average challenging behavior/task compliance, measured on a scale of 1-7 in which 1 is "Extremely Difficult" and 7 is "Exceptional" in the mattress technology on and off conditions
Time Frame: Average of daily measure, across up to 2 Weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Mattress Technology On | Mattress Technology Off
Number analyzed (Participants) | 45 | 45
units on a scale | 4.73 (0.12) | 4.35 (0.12)
Statistical Analysis 1: Comparison: Mattress Technology On vs Mattress Technology Off; Test type: Superiority; p = 0.001, Mixed Models Analysis

15. Secondary Outcome: Caregiver-Rated Measure of Tolerance of Mattress Technology as Measured by the Daily Sleep Diary
Description: Comparison of average tolerance of mattress technology, measured on a scale of 1-7 in which 1 is "Extremely Poor" and 7 is "Exceptional", in the on condition compared to the median score of 4 (average toleration of mattress technology).
Time Frame: Average of daily measure, across up to 2 Weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Mattress Technology On
Number analyzed (Participants) | 45
units on a scale | 5.61 (0.25)
Statistical Analysis 1: Comparison: Mattress Technology On; Test type: Non-Inferiority — Non-inferiority compared to the median rating of four on the seven point scale (1 = extremely poor, 7 = exceptional) that was used to rate tolerance; The mean rating of parent reported tolerance of mattress technology was 5.61 (SE = 0.25)

16. Secondary Outcome: Caregiver-Rated Measure of Tolerance of the Actigraph Watch as Measured by the Daily Sleep Diary
Description: Comparison of average tolerance of the actigraph watch, measured on a scale of 1-7 in which 1 is "Extremely Poor" and 7 is "Exceptional", across treatment conditions compared to median score of 4 (average toleration of actigraph watch).
Time Frame: Average of daily measure, across up to 4 Weeks
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- All Participants: All participants in both the mattress technology on and off conditions.
Arm/Group | All Participants
Number analyzed (Participants) | 45
units on a scale | 5.51 (0.13)
Statistical Analysis 1: Comparison: All Participants; Test type: Non-Inferiority — [test comment as in outcome 15, analysis 1]; The mean rating of parent reported tolerance of actigraph watch was 5.51 (SE = 0.13)

17. Secondary Outcome: Caregiver-Rated Measure of Ease of Mattress Technology Use as Measured by the Daily Sleep Diary
Description: Comparison of ease of mattress technology use, measured on a scale of 1-7 in which 1 is "Extremely Difficult" and 7 is "Exceptionally Easy" in mattress technology on condition to median score of 4 (average ease of use of mattress technology).
Time Frame: Average of daily measure, across up to 2 Weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Mattress Technology On
Number analyzed (Participants) | 45
units on a scale | 6.04 (0.15)
Statistical Analysis 1: Comparison: Mattress Technology On; Test type: Non-Inferiority — Non-inferiority compared to the median rating of four on the seven point scale (1 = extremely difficult, 7 = extremely easy) that was used to rate ease of use; The mean rating of parent reported ease of us of the mattress technology was 6.04 (SE = 0.15)

18. Secondary Outcome: Caregiver-Rated Measure of Sleep Resistance as Measured by the Daily Sleep Diary
Description: Within subjects comparison of average difficulty for child to go to bed, measured on a scale of 1-7 in which 1 is "Extremely Difficult" and 7 is "Exceptionally Easy", in the mattress technology on and off conditions.
Time Frame: Average daily measure, across up to 2 Weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Mattress Technology On | Mattress Technology Off
Number analyzed (Participants) | 23 | 22
units on a scale | 4.28 (0.14) | 4.79 (0.14)
Statistical Analysis 1: Comparison: Mattress Technology On vs Mattress Technology Off; Test type: Superiority; p = .001, Mixed Models Analysis; Mean Difference (Final Values) = 0.51

ADVERSE EVENTS:
Description: Same as Clinical Trials .Gov
Groups:
- Mattress Technology On: The mattress technology will be turned on.
  Intervention: The Sound to Sleep System is turned on allowing the participant sleeping atop the mattress to feel the vibrations synced to the audio input.
- Mattress Technology Off: The mattress technology is turned off, there is no intervention.
Arm/Group | Mattress Technology On | Mattress Technology Off
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 0/45 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No